CLINICAL TRIAL: NCT00306826
Title: Effect of Pioglitazone on Intima Media Thickness, Endothelial Function, and Heart Rate Variability in Patients With Impaired Glucose Tolerance
Brief Title: Pioglitazone in Impaired Glucose Tolerance
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: financial support withdrawn
Sponsor: University of Leipzig (Other)
Collaborators: Institut für Gesundheits- und Praxismanagement GmbH (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Leipzig-01
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2008-06

CONDITIONS: Glucose Metabolism Disorders
Keywords: Impaired glucose tolerance
MeSH Terms: conditions — Glucose Metabolism Disorders; Glucose Intolerance | interventions — Pioglitazone; Simvastatin

INTERVENTIONS:
Drug: pioglitazone
Drug: simvastatin
Drug: pioglitazone + simvastatin

SUMMARY:
In patients with impaired glucose tolerance (IGT), the researchers want to study the relative effects of pioglitazone, simvastatin, or the combination of both on:

* intima media thickness (IMT) as an easily assessed marker of atherosclerosis
* heart rate variability (HRV) as a marker of autonomic neuropathy
* flow-mediated vasodilatation (FMD) of the brachial artery as a marker of endothelial function
* vascular and metabolic lab parameters

DETAILED DESCRIPTION:
We want to study the relative effects of pioglitazone, simvastatin or the combination of both on intima media thickness (IMT), heart rate variability (HRV), flow-mediated vasodilatation (FMD) of the brachial artery and vascular/metabolic lab parameters in patients with impaired glucose tolerance (IGT). Previous studies have shown a reduction in IMT for both pioglitazone and simvastatin in type 2 diabetics. Many patients with diabetes mellitus develop diabetic polyneuropathy which can be assessed by measuring HRV. It has been shown that pioglitazone has a positive effect on HRV in type 2 diabetics. Questions remain on the relative efficacy of pioglitazone and simvastatin on the parameters mentioned above. Also, there is only scarce data in patients with IGT (as opposed to overt diabetes mellitus). There are no data on the relative effects of pioglitazone and simvastatin on flow-mediated vasodilatation (FMD) of the brachial artery as a surrogate marker for endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance
* Age 40 to 75 years

Exclusion Criteria:

* Diabetes mellitus type 1 or 2
* Hypersensitivity to study medication
* Malignant tumor
* Alcohol or drug abuse
* Overt heart failure
* Severe hepatic, renal, neurological, psychiatric, or hematological disease
* Prior treatment with glitazones or statins
* Established indication for statin treatment (e.g. coronary artery disease [CAD])

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Study Completion 2009-05

PRIMARY OUTCOMES:
Change in intima media thickness of carotid artery

SECONDARY OUTCOMES:
Heart rate variability
Flow-mediated dilatation of brachial artery
Vascular/metabolic lab parameters

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schuler, MD, Study Chair — University of Leipzig
Locations (7):
- Germany (7):
  - Praxis Antje Horn, Gera
  - Praxis Gunter Kässner, Leipzig
  - Praxis Heidrun Täschner, Leipzig
  - Praxis Martin Schönauer, Leipzig
  - University of Leipzig Heart Center, Leipzig
  - Praxis Matthias Weissbrodt, Leipzig
  - Praxis Matthias Schreiner, Leipzig

REFERENCES:
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751